CLINICAL TRIAL: NCT05333783
Title: Treating Cynophobia With Augmented Reality Exposure Therapy
Brief Title: Augmented Reality Exposure Therapy for Cynophobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022.034.IRB3.006
Record Dates: First submitted 2022-03-11; First posted 2022-04-19 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Phobia Animal
MeSH Terms: conditions — Zoophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Reality Exposure Therapy Based on ExposXR software (Experimental): The intervention arm will receive the assigned intervention in one session. Participants will be called for 2 times for post-assessment.
  Interventions: Behavioral: Augmented Reality Exposure Therapy Based on ExposXR software
- Treatment as Usual (No Intervention): The control arm has no intervention. However, the participants are not given any instruction limiting their encounters with the phobic stimuli. The participants in the control arm will receive the intervention after the post-assessments are completed.

INTERVENTIONS:
Behavioral: Augmented Reality Exposure Therapy Based on ExposXR software — The ExposXR software is developed by The Stress Trauma Anxiety Research Clinic at Wayne State University, U.S.A. When it is used inside a Augmented Reality hardware such as Hololens, it renders artificial phobic objects into what the participants see. The treatment consist of a one-session treatment for cynophobia using Augmented Reality.
  Arms: Augmented Reality Exposure Therapy Based on ExposXR software

SUMMARY:
The feasibility study for the Augmented Reality Exposure Therapy for Cynophobia will be carried out for people with dog phobia. This feasibility study's sample will be adults living in Turkey. The informed consent form and demographic form will be sent to the participants who have given this approval. Those who are eligible will be invited to diagnostic interviews. Those participants who meet the inclusion criteria will be included in the feasibility study. 22 participants are expected to participate in this study. The phobia severity will be measured three times: once before and twice after the intervention.

DETAILED DESCRIPTION:
Specific phobia is an overwhelming fear of an object, place, situation, feeling or animal. For the treatment of specific phobias, exposure therapy is accepted as the most effective way to treat the patients and it is frequently used by psychiatrists and psychotherapists. To treat specific phobias using exposure therapy, the patients are exposed to their feared objects or situations in a safe and controlled environment while they are guided and accompanied by a therapist. It is not always possible to conduct in vivo treatment however, due to a number of reasons such as the feared objects being unavailable, cost-effectiveness, patients with extremely high anxiety etc. Results of the former studies revealed that specific phobias can be treated using Augmented Reality (AR) where patients are exposed to virtually created feared objects in real life context. There are limited studies that have been conducted to test the effectiveness of AR because it is a newly developed technology. Former studies used AR to treat phobia of smaller object such as fear of cockroaches, insects and spiders. The current study aims to test whether AR is a successful tool that can be utilized as a treatment option for people with specific disorders. More specifically, we aim to test the effectiveness of Augmented Reality Exposure Therapy (ARET) in the treatment of patients with cynophobia, i.e., fear of dogs.

ELIGIBILITY:
Inclusion Criteria:

* Clinician-confirmed Dog Phobia
* Scoring 10 or higher on the Specific Phobia Scale (Adult version)

Exclusion Criteria:

* Psychosis and/or Substance Use Disorder
* Epileptic Seizure History
* Uncorrected Visual Impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Change of the Behavioral Approach Task (BAT) scores over time. | [Change from baseline (Before the intervention) to post assessment (1 week and 1 month after the pre-assessment) ]
  Specific Phobia Scale is a 10-item questionnaire that measures the severity of a specific phobia. Scores range from 0 (none) to 4 (severe).

SECONDARY OUTCOMES:
Change of the Specific Phobia Scale (SPS) Turkish version scores over time. | [Change from baseline (Before the intervention) to post assessment (1 week and 1 month after the pre-assessment) ]
  Specific Phobia Scale is a 10-item questionnaire that measures the severity of a specific phobia. Scores range from 0 (none) to 4 (severe).
Change of the Skin Conductance scores over time. | [Change from baseline (Before the intervention) to post assessment (1 week and 1 month after the pre-assessment) ]
  The skin conductance response, also known as the electrodermal response is the phenomenon that the skin momentarily becomes a better conductor of electricity when either external or internal stimuli occur that are physiologically arousing. Conductance is measured in μSiemens (μS) and is the inverse of electrical resistance.
Change of the Subjective Unit of Distress scores over time. | [Change from baseline (Before the intervention) to post assessment (1 week and 1 month after the pre-assessment) ]
  Subjective unit of distress (SUD) is a self-report measurement technique used to measure the intensity of distress or nervousness in people with anxiety. The SUDs are rated on a scale from 0 to 100. Higher scores indicate higher distress.

CONTACTS AND LOCATIONS:
Overall Officials: Can Anarat, MA, Study Chair — Koç University; Ekin Cakir, PhD, Study Chair — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Javanbakht A, Madaboosi S, Grasser LR. Real-life contextualization of exposure therapy using augmented reality: A pilot clinical trial of a novel treatment method. Ann Clin Psychiatry. 2021 Nov;33(4):220-231. doi: 10.12788/acp.0042. PMID 34672925

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT05333783/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT05333783/ICF_001.pdf